CLINICAL TRIAL: NCT03909191
Title: Serum HBV RNA Level Monitoring During Chronic Hepatitis B Virus Infection Especialy in Patients Undergoing Long-term Nucleos(t)Ide Analoguage Treatment
Brief Title: Serum HBV RNA Value on Chronic Hepatitis B Virus Infection Manage
Status: Completed | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, LiangXS, Associate professor, Changhai Hospital
Other Study IDs: HBV RNA2016
Record Dates: First submitted 2019-04-01; First posted 2019-04-09 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Chronic HBV Infection; Drug Withdrawal
Keywords: HBV RNA; HBsAg; cccDNA; Nucleos(t)ide analogue; virological relapse
MeSH Terms: conditions — Substance Withdrawal Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- treatment-naïve: treatment-naïve patients with chronic HBV infection
  Interventions: Diagnostic Test: serum HBV RNA
- NAs treated CHB patients: CHB patients undergoing long-term NAs treatment
  Interventions: Diagnostic Test: serum HBV RNA

INTERVENTIONS:
Diagnostic Test: serum HBV RNA — serum HBV RNA level was determined by using HBV-SAT kit at different time point

SUMMARY:
As an alternative biomarker of intrahepatic covalently closed circular DNA(cccDNA) transcriptional activity, hepatitis B virus(HBV)RNA may evolve during long-lasting virus-host interactionsduring chronic hepatitis B viral infection.The distribution pattern of serum HBV RNA levels in the natural course of chronic HBV infection remains unclear. Furthermore,serum HBV RNA was associated with response to NAs. So it may be another clinical surrogate marker for intrahepatic cccDNA level after long-term NAs treatment and be used to monitor NAs therapy. The aim of this study was to evaluate thelevels of HBV RNA during the natural courseof CHB and the role in distinguishingthe natural phases of HBV infection and to investigate whether serum HBV RNA level at the end of long-term NAs treatment had a similar or better predict effect on off-therapy relapse than serum HBsAg titer.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years old,
* no gender restriction,
* serum HBsAg positive than 6 months,
* can understand and sign informed consent,
* good compliance.

Exclusion Criteria:

* coinfected with other hepatotropic virus such as hepatitis C virus,hepatitis D -virus,hepatitis E and hepatitis A etc;
* coinfected with HIV,
* markers such as ceruloplasmin, anti-nuclear antibodies and anti-mitochondrial antibodies for co-existent autoimmune and metabolic liver diseases were positive,
* with hepatocellular carcinoma(HCC)
* with uncontrollable extrehepatic disease,
* received glucocorticoid or other immune inhibitor therapy,
* pregnancy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic Hepatitis B virus infection receiving or not receiving NAs treatment
Sampling Method: Non-Probability Sample
Enrollment: 454 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
serum HBV RNA value in treatment naive patients with chronic HBV infection were tested by using HBV SAT | serum HBV RNA level were measured 24hs after the enrollment
  serum HBV RNA level in patients with chronic HBV infection during different natural history stage were were compared. The relationship between serum HBV RNA and other viral markers,such as HBV DNA,HBeAg and HBsAg, were determined.
End of treatment serum HBV RNA levels predict the 24-month off-therapy viral rebound | Change in serum HBV DNA levels from stopping baseline to 24 month after drug cessation was determined
  End of treatment serum HBV RNA in patients after long-term nucleos(t)ide analog therapy were tested and the predictive effect of EOT HBV RNA value on 24-month off-therapy viral rebound were determined.

SECONDARY OUTCOMES:
serum HBV RNA in patients receiving long-term NAs therapy were tested at different time point | 48 hrs after enrollment the serun HBV RNA level were tested
  serum HBV RNA change pattern along long-term NAs therapy wad determined and the relationship between HBV RNA and HBV DNA or HBsAg during NAs therapy were also determined
Number of patients with evaluate HBV DNA relapse(> 20,000 IU/mL) through 96 weeks off-therapy | viral rebound rates were calculated from stopping baseline to 24 month after drug cessation
  the cumulative viral relapse rates at the 1st and 2nd year off-therapy were calculated

CONTACTS AND LOCATIONS:
Overall Officials: Xuesong Liang, Dr, Principal Investigator — Changhai Hospital

IPD SHARING:
Plan to Share IPD: No